CLINICAL TRIAL: NCT07043283
Title: A Phase I Study Evaluating the Single Subcutaneous Injection of Ebronucimab With Different Production Processes in Healthy Male Chinese Subjects
Brief Title: A Study Evaluating the Single Subcutaneous Injection of Ebronucimab in Healthy Male Chinese Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK102-103
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ebronucimab 150mg (after the change) (Experimental): Ebronucimab 150mg Single subcutaneous injection into the abdomen.
  Interventions: Drug: Ebronucimab
- Ebronucimab 150mg (before the change) (Experimental): Ebronucimab 150mg Single subcutaneous injection into the abdomen.
  Interventions: Drug: Ebronucimab

INTERVENTIONS:
Drug: Ebronucimab — Ebronucimab subcutaneous injection.

SUMMARY:
This is a phase I clinical study to evaluate the pharmacokinetics (PK) similarity of single dose subcutaneous injection of Ebronucimab with different production processes in Chinese healthy male subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel controlled, phase I clinical study to evaluate the pharmacokinetics (PK) similarity of single dose subcutaneous injection of Ebronucimab with different production processes in Chinese healthy male subjects. This study consists of two parts: pre-trial part and formal-trial part; with a planned sample size of 36 subjects in the pre-trial part, and 168 subjects in the formal trial part. A total of approximately 204 Chinese healthy male subjects are planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Subjects fully understand the purpose, content, process, and potential adverse events of the trial, voluntarily participate in the trial, and sign an informed consent form before any trial procedure begins.
* Weight: 60~80kg; Body mass index (BMI) ≥ 19 and ≤ 26 kg /m² for healthy Chinese male subjects.
* Fasting LDL-C level<4.1mmol/L.
* Fasting triglycerides<3.42mmol/L.
* Required to voluntarily adopt effective contraceptive measures as specified in the protocol throughout the entire trial period and within 3 months after receiving the investigational product, and avoid sperm donation.

Exclusion Criteria:

* 12 months prior use of PCSK9 inhibitors treatment.
* Allergic to the components of Ebronucimab and any monoclonal antibodies.
* History of important organ transplantation (such as heart, lung, liver, kidney, etc.).
* Abnormal vital signs during screening period and before randomization.
* Investigators believe that other factors may disqualify individuals from participating in the trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximum (peak) plasma concentration (Cmax) | Baseline till last follow-up visit (up to day 43 or day 57)
  Assess the Cmax of Ebronucimab.
Area under curve (AUC) | Baseline till last follow-up visit (up to day 43 or day 57)
  Assess the AUC of Ebronucimab.

SECONDARY OUTCOMES:
Incidence of adverse events (AE) | After the first administration till last follow-up visit (up to day 43 or day 57)
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Immunogenicity index | Day 1 and 43 ( or Day 57)
  Number and percentage of subjects with detectable anti drug antibodies (ADA) and neutralizing antibodies (Nab) after treatment.
Proprotein convertase subtilisin/kexin type 9 (PCSK-9) concentration | Day 1 and 43 ( or Day 57)
  Percentage change in PCSK-9 concentration compared to baseline.
Serum low-density lipoprotein cholesterol (LDL-C) concentration | Day 1 and 43 ( or Day 57)
  The change value and percentage of serum LDL-C concentration compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Xiaoshan Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No